CLINICAL TRIAL: NCT06611644
Title: A Comparative Analysis of Erector Spinae Plane (ESP) Block and Serratus Posterior Superior Intercostal Plane (SPSIP) Block in Breast Surgery
Brief Title: Comparison of ESP and SPSIP Blocks in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Mihrican SAYAN, Principal Investigator, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMU-SBF-ME-02
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Surgery; Macromastia; Mammaplasty; Modified Radical Mastectomy; Mammary Cancer; Breast Implant
Keywords: Pain Management; Regional Anesthesia; Multimodal Treatment; Modified Radical Mastectomy; Mammaplasty; Breast Implants
MeSH Terms: conditions — Gigantomastia; Breast Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: This study consists of three groups: a Control Group receiving standard postoperative pain management, an ESP Block Group receiving an Erector Spinae Plane (ESP) block, and an SPSIP Block Group receiving a Serratus Posterior Superior Intercostal Plane (SPSIP) block, all aimed at comparing the efficacy of these methods in managing postoperative pain.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be conducted in a double-blind design. Neither the patients nor the researchers assessing pain management will know which treatment has been applied. The anesthesia team, present in the operating room and responsible for administering the blocks, will be aware of the group assignments, but the research team responsible for postoperative evaluations will not have access to this information. The operating room coordinator will assign each patient to the appropriate group according to a randomization list and will only share this information with the anesthesia team. The research team evaluating postoperative pain scores and collecting data will do so without knowledge of the patients' treatment group, ensuring objectivity in the assessments through blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Erector Spinae Plane (ESP) block group (Active Comparator): This group will include patients who undergo the Erector Spinae Plane (ESP) block. The ESP block will be performed under ultrasound guidance, with a needle placed on the transverse process of the vertebra to inject local anesthetic into the erector spinae muscle.
  Interventions: Other: Erector Spinae Plane Block
- Serratus Posterior Superior Intercostal Plane (SPSIP) block (Active Comparator): This group will include patients who undergo the Serratus Posterior Superior Intercostal Plane (SPSIP) block. The SPSIP block will be performed under ultrasound guidance, injecting local anesthetic into the plane between the serratus posterior superior muscle and the intercostal muscles.
  Interventions: Other: SPSIPB blcok
- Control Group (Other): Patients in this group will receive standard postoperative pain management. This management will be provided through systemic analgesics (e.g., paracetamol, nonsteroidal anti-inflammatory drugs, and opioids if necessary) based on the patient's pain level during the postoperative period. This group will consist of patients who do not receive regional blocks, and pain management will be conducted according to the standard procedure of the surgery.
  Interventions: Other: Control

INTERVENTIONS:
Other: Erector Spinae Plane Block — Patients in this group will receive an Erector Spinae Plane (ESP) block in addition to standard postoperative care. The ESP block will be performed under ultrasound guidance. A needle will be advanced in-plane or out-of-plane, targeting the lateral aspect of the T6 transverse process. Local anesthetic (20 to 30 ml) will be injected into the fascial plane between the erector spinae muscle and the transverse process. This block is intended to provide postoperative analgesia by blocking the transmission of pain through the thoracic spinal nerves.
  Arms: Erector Spinae Plane (ESP) block group
Other: SPSIPB blcok — Patients in this group will receive a Serratus Posterior Superior Intercostal Plane (SPSIP) block along with standard postoperative care. The SPSIP block will be performed under ultrasound guidance, where the needle is advanced between the second and third ribs towards the medial aspect of the scapula. Local anesthetic 20 to 30 ml) will be injected into the fascial plane between the serratus posterior superior muscle and the intercostal muscles after confirming needle placement with hydrodissection using 1-2 ml of saline. This block is intended to provide broad analgesia across the upper thoracic dermatomes, from C3 to T7, to control postoperative pain.
  Arms: Serratus Posterior Superior Intercostal Plane (SPSIP) block
Other: Control — Patients in the control group will receive standard postoperative pain management without any regional block intervention. This will include the administration of systemic analgesics such as paracetamol and nonsteroidal anti-inflammatory drugs (NSAIDs). Opioid analgesics will be administered as needed based on the patient's pain level. Pain management will be conducted according to the standard protocol followed for breast surgery patients.
  Arms: Control Group

SUMMARY:
This study aims to compare the efficacy of the ESP and SPSIP blocks in managing postoperative pain following breast surgery. Breast surgery, particularly after oncological and reconstructive procedures, often leads to significant postoperative pain. Effective pain control is crucial for accelerating recovery, reducing the risk of complications, and facilitating early discharge. Both ESP and SPSIP blocks involve the administration of local anesthetics into fascial plane spaces to achieve peripheral nerve blockade and control pain. This study will evaluate the effectiveness of these blocks in terms of pain scores, opioid consumption, and overall patient satisfaction to determine the optimal approach for postoperative pain management in breast surgery.

DETAILED DESCRIPTION:
Breast surgery is one of the most frequently performed procedures, and effective postoperative pain management is critical to its success. Proper pain control not only facilitates early mobilization but also reduces the risks of pulmonary complications, deep vein thrombosis, and embolism. It helps prevent stress-induced endocrine and metabolic responses, shortens hospital stays, and lowers healthcare costs. Regional anesthesia is a highly effective strategy for postoperative pain control, minimizing opioid use and its associated side effects such as sedation, nausea, vomiting, and constipation.

Among the commonly used regional anesthesia techniques in breast surgery are the Erector Spinae Plane (ESP) block, Serratus Anterior Plane block, and Pectoral block. While the ESP block appears more effective, conflicting evidence exists regarding its efficacy in postoperative pain management, with variability in block spread across individuals. The recently introduced Serratus Posterior Superior Intercostal Plane (SPSIP) block, a periparavertebral block, offers a wider distribution range from C3 to T7 dermatomes, suggesting potential for more comprehensive postoperative analgesia in breast procedures.

The ESP block is performed under ultrasound guidance, using an in-plane technique to advance the needle from caudal to cranial (or vice versa), targeting the lateral part of the T6 transverse process, where local anesthetic is injected between the erector spinae muscle and the transverse process. For the SPSIP block, the needle is advanced between the second and third ribs towards the medial scapula, reaching the fascial plane between the serratus posterior superior muscle and the intercostal muscles. After hydrodissection confirms placement, local anesthetic is injected.

This study aims to compare the efficacy of ESP and SPSIP blocks in managing postoperative pain in breast surgery by evaluating pain scores, opioid consumption, and patient satisfaction. Since no study has yet directly compared these blocks, the findings will make a significant contribution to the existing literature.

ELIGIBILITY:
Inclusion Criteria

* Age between 18 and 65 years.
* Scheduled for breast surgery (Modified Radical Mastectomy with or without axillary lymph node dissection, Mastopexy, Reduction Mammoplasty).
* Preoperative anesthesia risk classified as ASA I-III according to the American -Society of Anesthesiologists (ASA) classification.
* Patients who provide informed consent for participation in the study.

Exclusion Criteria

* History of coagulation disorders.
* Patients using aspirin or medically prescribed anticoagulants.
* Patients with severe systemic diseases (ASA IV).
* Patients undergoing emergency surgery.
* Patients younger than 18 or older than 65 years.
* Patients who do not develop adequate sensory block after the procedure.
* Presence of infection at the block site.
* Patients with thoracic deformities.
* Patients who decline to participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals as female will be eligible to participate in this study, as the focus is on breast surgeries, which are performed on female patients.
Enrollment: 75 (Actual)
Dates: Start 2024-07-06 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Postoperative Opioid Consumption | 24 hours
  Postoperative opioid consumption will be monitored using a Patient-Controlled Analgesia (PCA) device, which will be connected to each patient at the end of surgery. The PCA settings will be 2 mg/cc tramadol solution, with no basal infusion, a lockout time of 20 minutes, and a 10 mg bolus dose. The total opioid (tramadol, Unit: miligram) consumption over 24 hours will be recorded, including the number of times the patient required analgesia and the number of bolus doses administered by the device.
Numeric Rating Scale (NRS) | 24 hours postoperatively (measured at 0, 2, 6, 12, and 24 hours)
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), where patients rate their pain on a scale from 0 (no pain) to 10 (worst possible pain). NRS scores will be recorded to evaluate postoperative pain levels in each group at specific intervals.

SECONDARY OUTCOMES:
Verbal Descriptive Nausea and Vomiting Scale | 24 hours postoperatively (measured at 0, 2, 6, 12, and 24 hours)
  Postoperative nausea and vomiting will be recorded for each patient at 0, 2, 6, 12, and 24 hours after surgery. The presence and severity of nausea and vomiting will be assessed using the Verbal Descriptive Nausea and Vomiting Scale, where 0 = none, 1 = mild nausea, 2 = moderate nausea, 3 = vomiting once, and 4 = vomiting more than once. This outcome will allow for a comparison of the potential of each technique to trigger postoperative nausea and vomiting.
Patient Satisfaction | 24 hours postoperatively
  Postoperative patient satisfaction will be measured to assess the overall acceptance and comfort related to the pain management strategies. Patient satisfaction will be rated on a three-point scale: good, moderate, or poor. This outcome will reflect the effectiveness of the pain management techniques in terms of patient comfort and overall experience.
Length of Hospital Stay | Up to 1 week postoperatively (measured in hours)
  The length of hospital stay (measured in hours) will be recorded for each patient to evaluate the potential for early discharge. A shorter hospital stay is typically associated with better pain management and faster recovery. This outcome will help assess the effectiveness of the pain control strategies in facilitating quicker recovery and discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No